CLINICAL TRIAL: NCT05460962
Title: Effects of Deep Breathing Excercises With and Without Progressive Muscle Relaxation Technique on Depression and Quality of Life in Females With Hystrectomy
Brief Title: Effects of Deep Breathing Excercises With and Without PMR on Depression & QOL in Females With Hystrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0515
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Post-Hysterectomy Vaginal Vault Prolapse
Keywords: Depression, Hysterectomy, Progressive muscle relaxation technique
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep breathing excercises (Experimental): is a technique that is based on the notion that mind and body integration produces relaxation technique requires participants to contract the diaphragm, slowly inhaling and exhaling. Deep breathing appears to amplify blood oxygen levels, massages the inner organs located in or close to the abdomen, and possibly stimulates the vagus nerve
  Interventions: Other: Deep breathing excercises; Other: Deep breathing exercises +and progressive muscle relaxation techniques
- Deep breathing excercise and progressive muscle relaxation (Experimental): Begin with a deep breathing exercise. Inhale deeply through your nose, feeling your abdomen rise as you fill your body with air. Then slowly exhale out the mouth, the navel pulling in toward the spine as you expel the stale air out. Repeat 3-5 cycles
  Interventions: Other: Deep breathing excercises; Other: Deep breathing exercises +and progressive muscle relaxation techniques

INTERVENTIONS:
Other: Deep breathing excercises — Deep breathing, which is also known as diaphragmatic breathing, is a technique that is based on the notion that mind and body integration produces relaxation technique requires participants to contract the diaphragm, slowly inhaling and exhaling. Deep breathing appears to amplify blood oxygen levels, massages the inner organs located in or close to the abdomen, and possibly stimulates the vagus nerve
Other: Deep breathing exercises +and progressive muscle relaxation techniques — Begin with a deep breathing exercise. Inhale deeply through your nose, feeling your abdomen rise as you fill your body with air. Then slowly exhale out the mouth, the navel pulling in toward the spine as you expel the stale air out. Repeat 3-5 cycles

SUMMARY:
To find out the Effects of deep breathing exercises with and without Progressive Muscle Relaxation Technique on depression and Quality of life in females with hysterotomy

ELIGIBILITY:
Inclusion Criteria:

* Age 35-55
* Females gone through all types of hysterotomy
* Hysterotomy done due to heavy menstrual bleeding, fibroids, pelvic pain, endometriosis and MAP ( Morbidly adherent placenta ).

Exclusion Criteria:

* Females with hormonal replacement therapy
* Any history of cancer
* Diagnosed patient of any psychiatric illness

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 8 weeks
  The Beck Depression Inventory (BDI) created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Its development marked a shift among mental health professionals, who had until then, viewed depression from a psychodynamic perspective, instead of it being rooted in the patient's own thoughts.
WHOQOL-BREFF | 8 weeks
  Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale (16, 17). The physical health domain includes items on mobility, daily activities, functional capacity, energy, pain, and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam Muneeb, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No